CLINICAL TRIAL: NCT07021222
Title: Multifactorial Strategies for the Prevention of the Risks of Ulceration in Patients Affected by Diabetic Foot
Brief Title: Multifactorial Strategies for the Prevention of the Risks of Ulceration in Patients Affected by Diabetic Foot (DARE-DiaFoot)
Acronym: DARE-DiaFoot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DARE-DiaFoot
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: population 1 will be enrolled with no previous history of foot ulceration, but has a moderate ulcerative risk (grade 2); population 2 is affected by diabetic foot, had foot ulcers (grade 3), but these must have been resolved from at least six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Population 1 (Other): Patients affected by diabetes mellitus type-2 with no previous history of foot ulceration, but with a moderate ulcerative risk.
  Interventions: Procedure: Full Analysis
- Population 2 (Other): Patients affected by diabetes mellitus type-2: typical adult subjects affected by diabetic foot, who had foot ulcers and thus in risk grade 3. The ulcerative lesions must have been resolved from at least 6 months, so that there is no longer acute inflammatory process in progress at the time of blood sampling.
  Interventions: Procedure: Partial Analysis

INTERVENTIONS:
Procedure: Full Analysis — Population 1 receives all three groups of analyses:Clinical-metabolical analyses, Biological-biochemical analyses, and Biomechanical-functional analyses.
  Arms: Population 1
Procedure: Partial Analysis — Population 2 receives two groups of analyses:Clinical-metabolical analyses and Biological-biochemical analyses.
  Arms: Population 2

SUMMARY:
This is a no-profit, multicentre, national, clinical trial for the prevention of the complications of the diabetic foot in two populations of patients with diabetes mellitus type-2.

DETAILED DESCRIPTION:
This is a no-profit, multicentre, national, clinical trial for the prevention of the complications of the diabetic foot in two populations of patients with diabetes mellitus type-2.

A first population has no previous history of foot ulceration, but has a moderate ulcerative risk (grade 2); a second population is affected by diabetic foot, had foot ulcers (grade 3), but these must have been resolved from at least six months.

One centre provides thorough biomechanical and functional analyses also based on modern Computed Tomography in weight-bearing; another centre performs state-of-the-art clinical assessments and metabolic analyses; the third centre performs the latter, together with advanced biological and biochemical analyses.

Comparisons of all these multi-instrumental measurements between the two populations are performed at baseline and at 12 month follow-up, with multidisciplinary investigative approach.

A mix of risk and predisposition factors should emerge combining the three groups of measures, in the two populations, along the two times of data collection.

ELIGIBILITY:
Inclusion Criteria for population 1:

* Male and female patients aged between 18 and 75 years.
* Diabetes mellitus type-2 patients with mild to moderate risk of ulceration at the foot (grade 2).

Inclusion Criteria for population 2:

* Male and female patients aged between 18 and 75 years.
* Patients with diabetes mellitus type-2 and diabetic foot with an history of ulcerative lesions (grade 3), healed for at least 6 months.

Exclusion Criteria for population 1:

* History or evidence of ulcers at the foot
* Infections in progress, ongoing neoplasms
* Immunosuppressive therapies, and cortisone-based therapy
* Pregnancy and lactation
* Inability to provide informed consent

Exclusion Criteria for population 2:

* Infections in progress, ongoing neoplasms
* Immunosuppressive therapies, and cortisone-based therapy
* Pregnancy and lactation
* Inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Biological biochemical analysis | baseline, 12 months
  Parameters related to the profile of blood biomarkers for inflammation will be acquired from samples collected for Population 1 and Population 2.

SECONDARY OUTCOMES:
Clinical - metabolical analysis | baseline, 12 months
  These evaluations will include the analysis of patients' medical history
Functional analysis | baseline, 12 months
  Instrumental evaluations are collected from only Population 1

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No
Data will not be shared until a full collection, analysis and major comprehension of the dataset by the scientists in the three centers involved; this dataset in fact is going to be very vast, very complex, and multi-disciplinary, and also the statistical analysis is expected to be difficult. These activities thus do deserve a careful scrutiny by the designers of the study before the dataset can be managed by other scientists; and this is going to take many years.

REFERENCES:
- [Background] van Netten JJ, Raspovic A, Lavery LA, Monteiro-Soares M, Paton J, Rasmussen A, Sacco ICN, Bus SA. Prevention of foot ulcers in persons with diabetes at risk of ulceration: A systematic review and meta-analysis. Diabetes Metab Res Rev. 2024 Mar;40(3):e3652. doi: 10.1002/dmrr.3652. Epub 2023 May 27. PMID 37243880
- [Background] Senneville E, Albalawi Z, van Asten SA, Abbas ZG, Allison G, Aragon-Sanchez J, Embil JM, Lavery LA, Alhasan M, Oz O, Uckay I, Urbancic-Rovan V, Xu ZR, Peters EJG. IWGDF/IDSA guidelines on the diagnosis and treatment of diabetes-related foot infections (IWGDF/IDSA 2023). Diabetes Metab Res Rev. 2024 Mar;40(3):e3687. doi: 10.1002/dmrr.3687. Epub 2023 Oct 1. PMID 37779323
- [Background] Leardini A, Benedetti MG, Berti L, Bettinelli D, Nativo R, Giannini S. Rear-foot, mid-foot and fore-foot motion during the stance phase of gait. Gait Posture. 2007 Mar;25(3):453-62. doi: 10.1016/j.gaitpost.2006.05.017. Epub 2006 Sep 11. PMID 16965916
- [Background] Ortolani M, Leardini A, Pavani C, Scicolone S, Girolami M, Bevoni R, Lullini G, Durante S, Berti L, Belvedere C. Angular and linear measurements of adult flexible flatfoot via weight-bearing CT scans and 3D bone reconstruction tools. Sci Rep. 2021 Aug 9;11(1):16139. doi: 10.1038/s41598-021-95708-x. PMID 34373546